CLINICAL TRIAL: NCT00748904
Title: A Randomized Comparison of Rifaximin Versus Lactulose in Hospitalized Cirrhotic Patients With Progressive Renal Failure
Brief Title: Rifaximin Versus Lactulose in Renal Failure
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0801009635
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Liver Cirrhosis; Renal Failure
Keywords: cirrhosis of liver and progressive renal failure
MeSH Terms: conditions — Liver Cirrhosis; Renal Insufficiency; Fibrosis | interventions — Rifaximin; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): 35 patients receiving rifaximin
  Interventions: Drug: Rifaximin
- B (Experimental): 35 patients receiving lactulose
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Rifaximin — 400 mg orally
  Other Names: Xifaxin, Salix Pharmaceuticals
  Arms: A
Drug: Lactulose — 20 grams titrate to 2-3 bowel movements in one day
  Arms: B

SUMMARY:
The purpose of this study is to evaluate patients with cirrhosis of the liver and renal failure and determine if the administration of rifaximin as compared to lactulose is associated with less frequent and/or slower progression to severe hepatic encephalopathy. If one is associated with lower blood ammonia levels. And, if one is associated with lower breath hydrogen and methane levels.

ELIGIBILITY:
Inclusion Criteria:

* cirrhosis of liver of any etiology
* progressive renal failure
* stage 0-2 hepatic encephalopathy

Exclusion Criteria:

* pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
slower progression to severe hepatic encephalopathy, stage 3 or 4 | during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States